CLINICAL TRIAL: NCT03889262
Title: Development of Simulated Hippotherapy System and Investigation of Its Effectiveness in Children With Cerebral Palsy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 09.2017.297
Record Dates: First submitted 2019-03-17; First posted 2019-03-26 (Actual); Last update posted 2019-03-28 (Actual); Status verified 2019-03

CONDITIONS: Cerebral Palsy
Keywords: Cerebral Palsy; Physiotherapy and Rehabilitation; Hippotherapy; Balance
MeSH Terms: conditions — Cerebral Palsy | interventions — Equine-Assisted Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): Participants in this group will receive only Neurodevelopmental therapy (NDT) based rehabilitation for 45 minutes in each session, twice a week, during 8 weeks, 16 sessions in total. Number of participants in this group is anticipated to be 20.
  Interventions: Other: Neurodevelopmental Therapy
- Study Group (Active Comparator): After 16 sessions (8 weeks) of only Neurodevelopmental therapy (NDT) based rehabilitation, simulated hippotherapy treatment will be added to rehabilitation program of the same participants. Their NDT treatment will be reduced to 25 minutes whereas hippotherapy will be applied for 20 minutes in each session, 2 sessions a week, 8 weeks in total.
  Interventions: Other: Hippotherapy; Other: Neurodevelopmental Therapy

INTERVENTIONS:
Other: Hippotherapy — Hippotherapy is a therapeutic method in which a mechanical horse is used for therapeutic purposes.
  Arms: Study Group
Other: Neurodevelopmental Therapy — Neurodevelopmental therapy (NDT) is a hands-on treatment approach used by physical therapists, occupational therapists, and speech-language pathologists. NDT was developed to enhance the function of children who have difficulty controlling movement as a result of neurological challenges, such as cerebral palsy and head injury. During treatment interventions, repeated experience in movement ensures that a particular pattern is readily accessible for motor performance. The more a patient performs certain movements, the easier these movements becomes.
  Other Names: Bobath Therapy

SUMMARY:
The purpose of this study is to develop a simulated hippotherapy system controlled by electromyography (EMG) signals and investigate its effectiveness in children with cerebral palsy. In order to investigate its effectiveness evaluation of gross motor functions, lower extremity joint movements, spasticity of the lower extremities, functional independence, body movements, sitting and standing balance, muscle tone, stiffness and elasticity level, analysis of the walking are planned.

DETAILED DESCRIPTION:
Hippotherapy is a therapeutic method in which a real horse is used for therapeutic purposes. It is widely used in many countries in the treatment of neuromuscular diseases (Multiple Sclerosis, stroke, Cerebral Palsy, etc.). Although the use of hippotherapy is widespread, many people can not reach and use this method effectively because of many reasons such as the high cost of caring, feeding, and sheltering horses or fear of people from horses. In recent years, hippotherapy simulation devices (mechanic and robotic horses) have been developed to overcome these problems. These devices aim to create the effects of hippotherapy on people by simulating a real horse's movement. The aim of this project is to develop and produce a simulated hippotherapy system, which can be controlled by electromyography (EMG) signals coming from the rider, movements programmable (for different musculoskeletal problems), rehabilitation-specific, providing evaluation during therapy, integrating virtual reality system and therapy games and investigate its effectiveness in children with cerebral palsy.

ELIGIBILITY:
Inclusion Criteria

* Having a diagnosis of Spastic Cerebral Palsy,
* Children aged between 5 - 18 years,
* Gross motor functional level is I, II or III,
* Independent seating
* Walking at least 10 meters independently,
* Can understand simple verbal instructions,
* Those with a spasticity level less than 2 according to Modified Ashworth Scale ,
* Having bilateral hip abduction enough to sit on the hippotherapy device,
* Voluntary acceptance to participate in the study

Exclusion Criteria

* Having hip dislocation,
* Severe contracture or deformity,
* Scoliosis (above 20 degrees),
* Acute uncontrolled acute seizures,
* Epilepsy,
* Visual and auditory problems,
* Injection of botulinum toxin in the last 6 months,
* History of surgical operation such as muscle relaxation, tendon extension and selective dorsal rhizotomy in the last 6 months.

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-04-01 (Estimated); Primary Completion 2019-09-20 (Estimated); Study Completion 2019-09-20 (Estimated)

PRIMARY OUTCOMES:
Change in functional level from baseline, week 8 and week 16 | 16 weeks
  Functional level will be defined with Gross Motor Functional Classification System (GMFCS). GMFCS defines movements such as sitting, walking and use of mobility devices. It provides a clear description of a child's current gross motor functional level. Level I can climb stairs without the use of a railing. Level II can walk in most settings and climb stairs holding onto a railing. Level III needs usage of a hand held mobility device, may climb stairs holding onto a railing with assistance. Level IV requires physical assistance or powered mobility in most settings. Level V children are transported in a manuel wheelchair in all settings, they are limited in their ability to maintain antigravity head and trunk postures and control leg and arm movements.
Change in spasticity from baseline, week 8 and week 16 | 16 weeks
  Spasticity will be defined with Modified Ashworth Scale (MAS). The MAS measures resistance during passive soft-tissue stretching. Scoring: 0= normal tone. 1= slight increase in muscle tone, minimal resistance at the end of the range of motion (ROM) when the affected part(s) is moved in flexion or extension. 1+= slight increase in muscle tone, manifested by a catch, followed by minimal resistance throughout the remainder of the ROM. 2= more marked increase in muscle tone through most of the ROM, but affected part(s) easily moved. 3= considerable increase in muscle tone, passive movement difficult. 4= affected part(s) rigid in flexion or extension.
Change in range of motion from baseline, week 8 and week 16 | 16 weeks
  Lower extremity Range of Motion (ROM) will be measured with universal goniometer.
Change in gross motor functional level from baseline, week 8 and week 16 | 16 weeks
  Gross motor function will be assessed with Gross Motor Function Measure-88. It consists of 88 items and contains 5 subdivisions: (A) reaching and turning; (B) sitting; (C) crawling and notebook; (D) standing; (E) walking, running and jumping. The total score and the scores of each sub-section are calculated. In our study, sections B, D and E will be evaluated.
Change in postural control from baseline, week 8 and week 16 | 16 weeks
  Trunk movements will be assessed with Trunk Impairment Scale (TIS). It will be used to evaluate the postural control. The scale is developed to evaluate the people with stroke and has been adapted and validated for the children with Cerebral Palsy (CP). The TIS assesses static and dynamic sitting balance and trunk coordination in a sitting position. The static subscale investigates the ability of the subject to maintain a sitting position with feet supported, while the legs are passively crossed, and when the subject crosses the legs actively. The dynamic subscale contains items on lateral flexion of the trunk and unilateral lifting of the hip. For each item, a 2, 3 or 4-point ordinal scale is used. On the static and dynamic sitting balance and coordination subscales the maximal scores that can be attained are 7, 10 and 6 points. The total score for TIS ranges between 0 for a minimal performance to 23 for a perfect performance.
Change in functional independence from baseline, week 8 and week 16 | 16 weeks
  Functional Independence will be defined with The Functional Independence Measure for Children (WeeFim). WeeFim consists of 6 parts: self-care, sphincter control, mobility, locomotion, communication and social communication. Each item is scored from 1 to 7 depending on whether it receives help when performing the function, whether it is on time, or whether the auxiliary device is required. "1" means fully dependent, "7" means fully independent. According to this, the highest score a child can get is 126 and the lowest score is 18.
Change in functional balance from baseline, week 8 and week 16 | 16 weeks
  Balance will be defined with Pediatrics Balance Scale (PDS). It is an assessment tool adapted from the Berg Balance Scale (BDS) to evaluate the functional balance of children in daily living activities. The scale consists of 14 chapters and each section is scored between 0 and 4; the highest score is 56. PDS is a high-reliability scale between groups and test re-testing in school-age children with mild to moderate motor impairment. The scale is valid in children with Cerebral Palsy.
Change in soft tissue from baseline, week 8 and week 16 | 16 weeks
  Soft tissue assessment will assessed with Myoton® PRO device. It is an evidence-based device that evaluates the bio-mechanical properties of soft biological tissues in a non-invasive, objective, reliable, inexpensive, quick and easy manner. Myoton® PRO is used in studies to evaluate superficial skeletal muscles, connective tissues such as tendons and ligaments, and other soft tissues. It is a highly reliable method for assessing the tone, stiffness, elasticity of muscles.
Change in walking from baseline, week 8 and week 16 | 16 weeks
  Walking analysis will be assessed with FreeMed® (Sensör Medica) which is a baropodometric platform. The software program can perform postural evaluation and bio-mechanical analysis. Dynamic analysis software program allows walking analysis. It documents the results in curves and graphics, podalic geometry, walking cycle, numerical values, combination of forces and videography and records in computer environment.
Change in body balance change from baseline, week 8 and week 16 | 16 weeks
  Balance will be assessed with Pedalo® Balance Device. It will be used to evaluate the balance during sitting and standing positions. Pedalo® balance device has been developed to record the user's movements to provide information about the body's balance, response time and possible imbalances. Pedalo® is a device that provides performance improvement in terms of balance and coordination. The device not only measures the performance that appears, but also compares previous performances to allow the evaluation of all performances.

CONTACTS AND LOCATIONS:
Overall Officials: Zubeyir Sarı, Study Director — Marmara University Institute of Health Sciences

IPD SHARING:
Plan to Share IPD: No
Study protocol, statistical analysis plan, informed consent form, clinical study report might be considered to be shared with the clinicians studying in the same field one year after the publication of the study.

REFERENCES:
- [Background] Champagne D, Corriveau H, Dugas C. Effect of Hippotherapy on Motor Proficiency and Function in Children with Cerebral Palsy Who Walk. Phys Occup Ther Pediatr. 2017 Feb;37(1):51-63. doi: 10.3109/01942638.2015.1129386. Epub 2016 Mar 1. PMID 26930110
- [Background] Han JY, Kim JM, Kim SK, Chung JS, Lee HC, Lim JK, Lee J, Park KY. Therapeutic effects of mechanical horseback riding on gait and balance ability in stroke patients. Ann Rehabil Med. 2012 Dec;36(6):762-9. doi: 10.5535/arm.2012.36.6.762. Epub 2012 Dec 28. PMID 23342307
- [Background] Herrero P, Gomez-Trullen EM, Asensio A, Garcia E, Casas R, Monserrat E, Pandyan A. Study of the therapeutic effects of a hippotherapy simulator in children with cerebral palsy: a stratified single-blind randomized controlled trial. Clin Rehabil. 2012 Dec;26(12):1105-13. doi: 10.1177/0269215512444633. Epub 2012 May 18. PMID 22610128
- [Background] Hosaka Y, Nagasaki M, Bajotto G, Shinomiya Y, Ozawa T, Sato Y. Effects of daily mechanical horseback riding on insulin sensitivity and resting metabolism in middle-aged type 2 diabetes mellitus patients. Nagoya J Med Sci. 2010 Aug;72(3-4):129-37. PMID 20942267
- [Background] Glanzman AM, Swenson AE, Kim H. Intrarater range of motion reliability in cerebral palsy: a comparison of assessment methods. Pediatr Phys Ther. 2008 Winter;20(4):369-72. doi: 10.1097/PEP.0b013e31818b7994. PMID 19011528
- [Background] Franjoine MR, Gunther JS, Taylor MJ. Pediatric balance scale: a modified version of the berg balance scale for the school-age child with mild to moderate motor impairment. Pediatr Phys Ther. 2003 Summer;15(2):114-28. doi: 10.1097/01.PEP.0000068117.48023.18. PMID 17057441
- [Background] Kim SG, Lee JH. The effects of horse riding simulation exercise on muscle activation and limits of stability in the elderly. Arch Gerontol Geriatr. 2015 Jan-Feb;60(1):62-5. doi: 10.1016/j.archger.2014.10.018. Epub 2014 Nov 7. PMID 25465508
- [Background] Kim SK, Kim SG, HwangBo G. The effect of horse-riding simulator exercise on the gait, muscle strength and muscle activation in elderly people with knee osteoarthritis. J Phys Ther Sci. 2017 Apr;29(4):693-696. doi: 10.1589/jpts.29.693. Epub 2017 Apr 20. PMID 28533611
- [Background] Kucukdeveci AA, Yavuzer G, Elhan AH, Sonel B, Tennant A. Adaptation of the Functional Independence Measure for use in Turkey. Clin Rehabil. 2001 Jun;15(3):311-9. doi: 10.1191/026921501676877265. PMID 11386402
- [Background] Lee CW, Kim SG, Na SS. The effects of hippotherapy and a horse riding simulator on the balance of children with cerebral palsy. J Phys Ther Sci. 2014 Mar;26(3):423-5. doi: 10.1589/jpts.26.423. Epub 2014 Mar 25. PMID 24707098
- [Background] Lee DR, Lee NG, Cha HJ, Yun Sung O, You SJ, Oh JH, Bang HS. The effect of robo-horseback riding therapy on spinal alignment and associated muscle size in MRI for a child with neuromuscular scoliosis: an experimenter-blind study. NeuroRehabilitation. 2011;29(1):23-7. doi: 10.3233/NRE-2011-0673. PMID 21876292
- [Background] Lee J, Yun CK. Effects of hippotherapy on the thickness of deep abdominal muscles and activity of daily living in children with intellectual disabilities. J Phys Ther Sci. 2017 Apr;29(4):779-782. doi: 10.1589/jpts.29.779. Epub 2017 Apr 20. PMID 28533630
- [Background] Leveille A, Rochette A, Mainville C. Perceived risks and benefits of hippotherapy among parents of children currently engaged in or waiting for hippotherapy: A pilot study. Physiother Theory Pract. 2017 Apr;33(4):269-277. doi: 10.1080/09593985.2017.1302029. Epub 2017 Apr 5. PMID 28379061
- [Background] Mutlu A, Livanelioglu A, Gunel MK. Reliability of goniometric measurements in children with spastic cerebral palsy. Med Sci Monit. 2007 Jul;13(7):CR323-9. PMID 17599027
- [Background] Mutlu A, Livanelioglu A, Gunel MK. Reliability of Ashworth and Modified Ashworth scales in children with spastic cerebral palsy. BMC Musculoskelet Disord. 2008 Apr 10;9:44. doi: 10.1186/1471-2474-9-44. PMID 18402701
- [Background] Palisano R, Rosenbaum P, Walter S, Russell D, Wood E, Galuppi B. Development and reliability of a system to classify gross motor function in children with cerebral palsy. Dev Med Child Neurol. 1997 Apr;39(4):214-23. doi: 10.1111/j.1469-8749.1997.tb07414.x. PMID 9183258
- [Background] Park JH, Shurtleff T, Engsberg J, Rafferty S, You JY, You IY, You SH. Comparison between the robo-horse and real horse movements for hippotherapy. Biomed Mater Eng. 2014;24(6):2603-10. doi: 10.3233/BME-141076. PMID 25226963
- [Background] Saether R, Helbostad JL, Adde L, Jorgensen L, Vik T. Reliability and validity of the Trunk Impairment Scale in children and adolescents with cerebral palsy. Res Dev Disabil. 2013 Jul;34(7):2075-84. doi: 10.1016/j.ridd.2013.03.029. Epub 2013 May 1. PMID 23643761
- [Background] Silva e Borges MB, Werneck MJ, da Silva Mde L, Gandolfi L, Pratesi R. Therapeutic effects of a horse riding simulator in children with cerebral palsy. Arq Neuropsiquiatr. 2011 Oct;69(5):799-804. doi: 10.1590/s0004-282x2011000600014. PMID 22042184
- [Background] Yi SH, Hwang JH, Kim SJ, Kwon JY. Validity of pediatric balance scales in children with spastic cerebral palsy. Neuropediatrics. 2012 Dec;43(6):307-13. doi: 10.1055/s-0032-1327774. Epub 2012 Sep 25. PMID 23011753

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2019-02-28): https://cdn.clinicaltrials.gov/large-docs/62/NCT03889262/Prot_SAP_ICF_000.pdf